CLINICAL TRIAL: NCT07137806
Title: Beyond the Joint: Enhanced Pain Relief With Ultrasound Guided Combined Submaltifidus and Sacroiliac Joint Injection - a Randomized Controlled Trial
Brief Title: Enhanced Pain Relief With Ultrasound Guided Combined Submaltifidus and Sacroiliac Joint Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mohamed Shebl Abdelghany (Unknown)
Responsible Party: Principal Investigator, Aliaa Muhammad Belal, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Faculty of Medicine, Tanta Uni
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound guided sacroiliac joint injection group (Active Comparator): patients included in this group will receive SIJ injection alone.The injectate includes 40 mg of methylprednisolone acetate diluted in 2 mL of bupivacaine 0.25% with epinephrine 1:200,000 (total 3 mL injectate).
  Interventions: Procedure: sacroiliac joint injection
- combined ultrasound guide sacroiliac joint injection and submaltifidous plan (combined block group): (Experimental): patients included in this group will receive combined SMPB and SIJ injection twenty millilitres of local anaesthetic solution (1:1 mixture of lidocaine 2% and bupivacaine 0.25%) will be injected in the plane between the multifidus muscle (MFM) and the hyperechoic bony area (between the median and intermediate sacral crests)
  Interventions: Procedure: combined sacroiliac joint injection and sub maltifidous plane block

INTERVENTIONS:
Procedure: sacroiliac joint injection — Ultrasound-guided injection of the SI joints The patient is placed in a prone position to receive this injection treatment. The Curvilinear transducer is placed in a transverse orientation to identify the sacral hiatus first. After identifying the sacral cornu, the transducer is moved in a lateral direction until the lateral edge of the sacrum is observed. With the transducer maintained in the transverse orientation, it is then moved in a cephalad or upward direction until the bony contour of the ileum is identified. The cleft between the bony contours of the sacrum and ileum represents the posterior aspect of the SI joint. By tilting the transducer in a caudal direction, the lower one third of the SI joint is identified. Because of its synovial component, the lower one third of the SI joint is the portion of the entire SI joint in which the injection should be performed. The medial to lateral approach and intraarticular deposition is preferred for the ultrasound-guided SI joint
  Arms: ultrasound guided sacroiliac joint injection group
Procedure: combined sacroiliac joint injection and sub maltifidous plane block — patients will be positioned prone. A 6-13 MHz linear array ultrasound transducer was placed in the parasagittal orientation with the second sacral foramen (SF-2) in the field. A 21G short bevel needle is inserted in-plane approach from the cephalad to the caudad direction. After hitting the underlying bone, twenty millilitres of local anaesthetic solution (1:1 mixture of lidocaine 2% and bupivacaine 0.25%) will be injected. An anechoic LA spread in the plane between the multifidus muscle (MFM) and the hyperechoic bony area (between the median and intermediate sacral crests) will be confirmed. The Curvilinear transducer is placed in a transverse orientation to identify the sacral hiatus first. After identifying the sacral cornu, the transducer is moved in a lateral direction until the lateral edge of the sacrum is observed. With the transducer maintained in the transverse orientation, it is then moved in a cephalad or upward direction until the bony contour of the ileum is identified.
  Arms: combined ultrasound guide sacroiliac joint injection and submaltifidous plan (combined block group):

SUMMARY:
Sacroiliitis is not the same as SI joint dysfunction. Sacroiliitis is specific to an inflammatory processes present in the SI joint and the pain sensed is a direct result of those inflammatory processes, whereas sacroiliac joint dysfunction is a condition caused by abnormal motion or slight mispositioning of the SI joint.

Sacroiliac joint syndrome is a condition that is difficult to diagnose and is often overlooked by physicians and physiotherapist

DETAILED DESCRIPTION:
Treatment of SI joint pain usually involves a multi-pronged approach, utilizing both, multi-modal medical pain control and interventional pain/surgical techniques such as local anesthetic and steroid injections, radiofrequency nerve ablation, and minimally invasive sacroiliac arthrodesis.[7] Sacroiliac (SI) joint injection is a minimally invasive procedure that involves injecting a mixture of local anesthetic and/or corticosteroid medication directly into the SI joint[8] Depending on the mixture of medications used, the duration of pain relief varies but can last anywhere from several days to months[9] Local anesthetic and corticosteroid medications are used to reduce inflammation and provide symptom relief to patients with arthritis, inflammatory conditions, and/or acute injuries[10]

The goal of SI joint injections is to provide enough pain relief to allow the patient to improve their functional status. Participation in physical therapy or exercise is encouraged, which can lead to longer-term improvements in pain and function. The number of SI joint injections required for effective pain relief can vary depending on the patient. [11, 12] Some patients may only require one injection, while others may require several injections. As a general guideline, injections may be administered once every 2 weeks, and no more than 3 injections may be given per year[11, 12] In general, if the first injection provides significant relief, additional injections may be recommended. However, the exact timing can vary based on the doctor's guidance, the patient's response to the treatment, and the type of injection[13] The long-term outcomes of SI joint injections can vary depending on a number of factors, including the underlying cause of the pain, the patient's overall health, the patient's response to the injection, and the type of injection used. Steroid injections may work well for some patients, while others may respond more positively to prolotherapy or PRP therapy[14]

Sacral Multifidus Plane Block(SMPB), a variant of paraspinal plane blocks, has been used for various surgeries in the perineal and buttock region[15]

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 21 years, both genders diagnosed with chronic sacroiliac joint pain with a rating on the numeric pain rating scale (NPRS) of at least 5, without radiculopathy lasting 3 months or longer, and lack of medical treatment satisfactory response

Exclusion Criteria:

Patient refusal. Patients who have any allergies to local anesthetics or have had a reaction to contrast dyes in the past.

Patients who are unable to describe their pain (e.g., language barrier or neuropsychiatric disorder).

Patients with history of bleeding diathesis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Sacroiliac joint pain assessment according to Numerical rating Scale at 1month after injection. | at one month from intervention

SECONDARY OUTCOMES:
Analgesics consumption during 6month follow-up period | over 6 month from intection
Level of disability was measured by Oswestry Disability Index (ODI) scores | 6 month after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
individual issues